CLINICAL TRIAL: NCT04998188
Title: Hydrolyzed Collagen Formulation Versus Placebo in the Treatment of Degenerative Knee Cartilage Injuries
Brief Title: Hydrolyzed Collagen Formulation vs Placebo in Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: COLL-OA
Record Dates: First submitted 2021-05-17; First posted 2021-08-10 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee; knee osteoarthritis; collagen; collagen injection; osteoarthritis; placebo; Randomized controlled trial; double-blinded
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Collagen; Saline Solution

STUDY DESIGN:
Intervention Model Description: The study is a double-blinded RCT with possibility ,after 6 months, to cross-over from control arm (saline solution ) to the treatment arm (collagen). After 6 months, patients in the control arm have the possibility to cross-over into the treatment arm, in which case they will be followed for an additional 6 months
Who Masked: Participant, Outcomes Assessor
Masking Description: his is a double-blind randomized controlled trial with 1:1 allocation. Patients, healthcare professionals who assess clinical and functional outcomes (outcome assessors) and professionals who analyze the data will be "blinded."
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collagen Injection (Experimental): This group of patients will be treated with single intra-articular injection of collagen.
  Interventions: Procedure: Collagen
- Placebo (saline solution) (Placebo Comparator): This group of patients will be treated with single intra-articular injection of saline solution (placebo). At the 6-month follow-up visit, patients will be informed about the treatment received. Patients of this group can cross-over to the treatment arm after 6 months.
  Interventions: Procedure: Placebo (saline solution)

INTERVENTIONS:
Procedure: Collagen — Patients will be treated with a single injection of collagen (2 ml) in the knee joint affected by osteoarthritis
  Arms: Collagen Injection
Procedure: Placebo (saline solution) — Patients will be treated with a single injections of saline solution (2 ml) in the knee joint affected by osteoarthritis
  Arms: Placebo (saline solution)

SUMMARY:
The aim of the study is to compare the 6 months clinical outcome of the treatment with a single intra-articular collagen injection versus a single placebo (saline solution) infiltration in the infiltrative treatment of knee osteoarthritis. The evaluation will be performed through clinical, subjective and objective assessments.

DETAILED DESCRIPTION:
204 patients affected by knee osteoarthritis will be included in a double-blinded randomized controlled trial. Patients in the experimental group will be treated with a single intra-articular injection of collagen (solution of low molecular weight peptides derived from hydrolyzed collagen) instead patients in the control arm, will be treated with a single intra-articular injection of placebo (saline solution). All patients will be evaluated by clinical examination before the infiltrative procedure and they will follow-up at 1,3,6 months. During the follow-up visits ,will be evaluated the inflammatory status of the knee by thermographic assessment and questionnaires, filled out by patients, will be utilized for clinical evaluations. After 6 months, patients in the control arm (saline solution injection), have the possibility to cross-over into the treatment arm (collagen) in which case they will be followed for an additional 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral involvement;
2. Signs and symptoms of degenerative pathology of knee cartilage;
3. Radiographic and MRI signs of degenerative pathology of the knee cartilage (Kellgren-Lawrence 1-4 grades);
4. Failure, defined as the persistence of symptoms, after at least one course of conservative treatment (pharmacological, physiotherapeutic or infiltrative treatment);
5. Ability and consent of patients to actively participate in clinical follow-up;

Exclusion Criteria:

1. Patients who have undergone intra-articular injections of another substance in the previous 6 months;
2. Patients undergoing knee surgery within the previous 12 months;
3. Patients with malignant neoplasms;
4. Patients with rheumatic diseases;
5. Patients with diabetes;
6. Patients with hematologic diseases (coagulopathies);
7. Patients on anticoagulant therapy;
8. Patients with metabolic disorders of the thyroid gland;
9. Patients abusing alcoholic beverages, drugs or medications;
10. Body Mass Index > 35;
11. Pregnant or lactating women.
12. Patients with established hypersensitivity to bovine collagen or vitamin C.
13. Patients with joint or peri-articular infections, emarto, erythema, or psoriatic patches in the knee joint area

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 204 (Estimated)
Dates: Start 2022-02-16 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
KOOS-Pain Score | 6 months follow-up
  KOOS-Pain Score is referred to a subscale of pain composed by 9 items. The score range considerate is 0-100.The score uses a 5-point Likert scale and each question is assigned a score from 0 to 4, where 0 indicates "no pain" and 4 "severe level of pain"

SECONDARY OUTCOMES:
IKDC-Subjective Score | baseline, 1 month, 3 months, 6 months follow-up
  This is a subjective, knee-specific rating scale that is considered one of the most reliable assessment tools in the evaluation of knee pathologies. All questions examines 3 categories: symptoms, sports activity, and knee function
KOOS Score | baseline, 1 month, 3 months, 6 months follow-up
  KOOS SCORE consists of 5 subscales and covers: pain (9 items), symptoms (7 items, two of which are related to stiffness), functions and activities of daily living (17 items), physical function, sports and leisure activities (5 items) and quality of life in relation to the knee (4 items).
  Each question is scored from 0 to 4, where 0 indicates "no difficulty" and 4 "severe difficulty. Score range 0-100 for each subscale
WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) score | baseline, 1 month, 3 months, 6 and 12 months follow-up
  It's a standardized questionnaire to assess the condition of patients affected by knee osteoarthritis and includes assessment of pain, stiffness and physical functioning of the joints. It measures 5 items for pain (range 0-20), two for stiffness (range 0-8) and 17 for functional limitation (range 0-68) that relate mainly to activities of daily living. The score is normalized on a 0-100 scale. Higher values indicate a worse outcome.
VAS-pain (Visual Analogue Scale) | baseline, 1 month, 3 months, 6 months follow-up
  VAS is a visual analogue scale consisting of a range scale (10 cm length), the ends of which correspond to "no pain" and "the strongest pain imaginable".
EQ-VAS | baseline, 1 month, 3 months, 6 months follow-up
  EQ-VAS Is a visual analog scale that has a range of scores from 0 (worst imaginable health condition) to 100 (best imaginable health condition).
EQ-5D (EuroQoL) Current Health Assessment | baseline, 1 month, 3 months, 6 months follow-up
  The EQ-5D profile, asks patients to classify their health based on self-assessed levels of problems ("no", "some", "extreme") on five dimensions.
TegnerActivity Level Scale | baseline, 1 month, 3 months, 6 months follow-up
  Tegner activity level scale allows to know the level of physical activity carried out by the patients. Tegner's activity scale classifies the activity according to work and sports activities on a scale from 0 to 10. Zero represents disability because of knee problems and 10 represents soccer a national or international level
Patient Acceptable Symptom State (PASS) | baseline, 1 month, 3 months, 6 months follow-up
  A tool to assess patient satisfaction in consideration of their current degree of pain, function, and daily activity. Patients can express if their state of health will be satisfying, answering "yes" or "no".
Objective parameters -Range of motion | baseline, 1 month, 3 months, 6 months follow-up
  Evaluation of the Range of Motion for comparative analysis.
Final treatment opinion | 6 months follow-up
  The patient should indicate satisfaction and relative degree with treatment at the end of the clinical trial (24 months follow-up). All patients will be able to indicate their health condition by choosing from this answers; "Full recovery", "much better", "somewhat better", "no change", "a little worse", "much worse".
Ultrasound assessment | Baseline
  This examination is useful to do an initial assessment of possible meniscal extrusion in the interested knee joint.
Thermographic evaluation of the inflammatory status of the knee joint | baseline, 1 month, 3 months, 6 months follow-up
  The evaluation will be performed through the use of a thermal imaging camera. The thermal camera will allow to detect even small variation of knee temperature thus comparing and recording any thermographic changes in the inflammatory state of the joint before and after treatment.
Objective parameters - Circumferences | baseline, 1 month, 3 months, 6 months follow-up
  Bilateral trans- and supra- patellar circumferences measurement for comparative analysis

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Di Martino, MD, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Filardo G, Kon E, Longo UG, Madry H, Marchettini P, Marmotti A, Van Assche D, Zanon G, Peretti GM. Non-surgical treatments for the management of early osteoarthritis. Knee Surg Sports Traumatol Arthrosc. 2016 Jun;24(6):1775-85. doi: 10.1007/s00167-016-4089-y. Epub 2016 Apr 4. PMID 27043347
- [Background] Volpi P, Zini R, Erschbaumer F, Beggio M, Busilacchi A, Carimati G. Effectiveness of a novel hydrolyzed collagen formulation in treating patients with symptomatic knee osteoarthritis: a multicentric retrospective clinical study. Int Orthop. 2021 Feb;45(2):375-380. doi: 10.1007/s00264-020-04616-8. Epub 2020 May 23. PMID 32447428
- [Background] De Luca P, Colombini A, Carimati G, Beggio M, de Girolamo L, Volpi P. Intra-Articular Injection of Hydrolyzed Collagen to Treat Symptoms of Knee Osteoarthritis. A Functional In Vitro Investigation and a Pilot Retrospective Clinical Study. J Clin Med. 2019 Jul 4;8(7):975. doi: 10.3390/jcm8070975. PMID 31277508
- [Background] Farr J, Gomoll AH, Yanke AB, Strauss EJ, Mowry KC; ASA Study Group. A Randomized Controlled Single-Blind Study Demonstrating Superiority of Amniotic Suspension Allograft Injection Over Hyaluronic Acid and Saline Control for Modification of Knee Osteoarthritis Symptoms. J Knee Surg. 2019 Nov;32(11):1143-1154. doi: 10.1055/s-0039-1696672. Epub 2019 Sep 18. Erratum In: J Knee Surg. 2019 Nov;32(11):e2. doi: 10.1055/s-0039-3402742. PMID 31533151
- [Background] Furuzawa-Carballeda J, Munoz-Chable OA, Barrios-Payan J, Hernandez-Pando R. Effect of polymerized-type I collagen in knee osteoarthritis. I. In vitro study. Eur J Clin Invest. 2009 Jul;39(7):591-7. doi: 10.1111/j.1365-2362.2009.02154.x. PMID 19453649
- [Background] Vucic K, Jelicic Kadic A, Puljak L. Survey of Cochrane protocols found methods for data extraction from figures not mentioned or unclear. J Clin Epidemiol. 2015 Oct;68(10):1161-4. doi: 10.1016/j.jclinepi.2014.11.016. Epub 2014 Dec 18. PMID 25577327